CLINICAL TRIAL: NCT00691977
Title: A Phase I Dose-Escalation Study of Preoperative Radiation Therapy Followed by Radical Prostatectomy in Patients With High-Risk, Localized Carcinoma of the Prostate
Brief Title: Radiation Therapy Followed by Surgery in High-Risk, Localized Carcinoma of the Prostate
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Duke-10571
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: Radiation Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Radiation Therapy followed by prostatectomy
  Interventions: Radiation: Radiation Therapy followed by prostatectomy

INTERVENTIONS:
Radiation: Radiation Therapy followed by prostatectomy — Radiation Therapy

SUMMARY:
The purpose of the study is to assess the safety of four different doses of radiation therapy followed by to surgery to remove prostate tumor.

DETAILED DESCRIPTION:
Patients in Groups 1 and 2 will receive 39.6 Gy and 45 Gy (at 1.8 Gy/fraction), respectively, to the whole pelvis. Patients in Groups 3 and 4 will receive 45 Gy to the whole pelvis, followed by a boost to the prostate and periprostatic tissue, for total doses of 50.4 and 54 Gy, respectively. The patients will then undergo radical prostatectomy between 4-8 weeks after completion of radiation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have biopsy-confirmed adenocarcinoma of the prostate.
* Subjects must have a negative bone scan.
* Subjects must have "high-risk" prostate cancer, defined as:

A. PSA >/= 20, and/or B. Gleason Score (GS) >/= 8, and/or C. Clinical stage T3 disease per AJCC Staging Manual, 6th edition; or D. At least two out of three of the following: PSA 10-19.9, GS = 7, or clinical stage = T2b / T2c.

* Subjects must be medically fit to undergo surgery as determined by treating urologist.
* Subjects must be under 70 years of age.
* KPS must be >/= 80.
* Subjects must not have a synchronous primary tumor, or a previous cancer unless disease free for >/= 5 years.
* Subjects must not have had prior pelvic radiation therapy, chemotherapy, or androgen deprivation.
* Subjects must freely sign informed consent to enroll in the study.

Exclusion Criteria:

* Metastatic disease as demonstrated by bone scan, CT scan or MRI of the pelvis, or chest x-ray.
* Pathologically documented positive pelvic lymph nodes. If Pre-operative CT scan or MRI (ordered at the discretion of the treating physicians) demonstrates lymph nodes which are suspicious for involvement, then biopsy must be undertaken and nodes proven negative before patient can enroll on this trial.
* Declared high-risk for anesthesia by attending anesthesiologist, cardiologist, or other physician.
* History of prior pelvic radiation therapy.
* History of androgen deprivation therapy or chemotherapy.

Max Age: 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluate number of patients who are able to undergo surgery after preoperative radiation therapy. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S. Anscher, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States